CLINICAL TRIAL: NCT01100489
Title: A Phase II Study of the Feasibility and Efficacy of Breast Conserving Surgery in Patients With MRI Detected Multi-Centric Breast Cancer
Brief Title: Breast-Conserving Surgery Followed by Radiation Therapy With MRI-Detected Stage I or Stage II Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1109; NCI-2010-00644 (Other: NCI/CTRP)
Record Dates: First submitted 2010-04-07; First posted 2010-04-09 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Ductal Breast Carcinoma in Situ; Estrogen Receptor-negative Breast Cancer; Estrogen Receptor-positive Breast Cancer; HER2-negative Breast Cancer; HER2-positive Breast Cancer; Invasive Ductal Breast Carcinoma; Invasive Lobular Breast Carcinoma; Male Breast Cancer; Medullary Ductal Breast Carcinoma With Lymphocytic Infiltrate; Mucinous Ductal Breast Carcinoma; Papillary Ductal Breast Carcinoma; Progesterone Receptor-negative Breast Cancer; Progesterone Receptor-positive Breast Cancer; Stage I Breast Cancer; Stage II Breast Cancer; Tubular Ductal Breast Carcinoma
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Carcinoma, Ductal, Breast; Carcinoma, Lobular; Breast Neoplasms, Male; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients undergo breast-conserving surgery consisting of partial mastectomies followed by external beam breast radiation therapy 5 days a week for 5 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: external beam radiation therapy; Other: questionnaire administration; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Radiation: external beam radiation therapy — External beam breast radiation therapy 5 days a week for 5 weeks in the absence of disease progression or unacceptable toxicity.
  Other Names: EBRT
Other: questionnaire administration — Ancillary studies: The patient will complete the Cosmesis /QOL form (Appendix II) and the treating physician will complete the Cosmetic Guidelines (skin assessment) form for baseline data (Appendix I).
Procedure: therapeutic conventional surgery — Patients will undergo excisional biopsy or needle localization removal of the tumor. Patients with margins < 2 mm undergo re-excision of the biopsy cavity. Surgical clips should be placed at the time of tylectomy to define the excision cavities. Ideally, clips are to be placed marking the superficial, deep, right, left, inferior, and superior dimensions of the tylectomy or re-excision cavities.

SUMMARY:
RATIONALE: Breast-conserving surgery is a less invasive type of surgery for breast cancer and may have fewer side effects and improve recovery. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving radiation therapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II clinical trial is studying how well breast-conserving surgery followed by radiation therapy works in treating patients with stage I or stage II breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine ipsilateral breast tumor recurrence rates as well as tumor bed recurrence rates. Patients will be followed for a period of five years following completion of radiation to determine these rates.

II. To determine the cosmetic outcome resulting from breast conserving surgery and breast radiation.

SECONDARY OBJECTIVES:

I. To determine if there are patient factors which limit a patient's suitability to receive breast conserving therapy in the setting of multi-centric disease.

II. To determine patient satisfaction of breast conserving therapy as it pertains to their overall treatment experience as measured by a questionnaire.

III. To evaluate wound healing and overall complication rate after radiation as a component of breast conserving therapy.

OUTLINE:

Patients undergo breast-conserving surgery consisting of partial mastectomies followed by external beam breast radiation therapy 5 days a week for 5 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 1 month, then every 3 months for 1 year, every 6 months for 1 year, and then annually for 5 years.

ELIGIBILITY:
Inclusion

* Patients with multicentric carcinoma (tumors in different quadrants of the breast or tumors separated by at least 4 cm)
* All radiographically suspicious lesions must be biopsied and have histologically confirmed ductal carcinoma in-situ, invasive ductal, invasive lobular, medullary, papillary, colloid (mucinous), or tubular histologies
* A maximum of two radiographically detected malignant lesions
* Clinical Stage I-II breast carcinoma, with lesion size =< 5 cm for the dominant mass and the second lesion detected only on MRI, treated with lumpectomies; the MRI detected lesion must be pathologically =< 1 cm
* Axillary lymph node evaluation, either sentinel lymph node biopsy or axillary dissection as deemed appropriate by the treating surgeon for all patients with invasive cancer; no axillary lymph node sampling is needed for patients with DCIS
* Negative resection margins with at least a 2 mm margin from invasive and in-situ cancer or a negative re-excision
* A posterior margin =< 2 mm from DCIS is permissible provided fascia was taken
* Patients are eligible regardless of estrogen receptor, progesterone receptor, or Her-2/neu amplification
* Hormonal therapy is allowed; if adjuvant chemotherapy is planned, the chemotherapy should be delivered first and radiation must begin no earlier than three weeks and no later than eight weeks following completion of chemotherapy
* Signed study-specific informed consent prior to study entry

Exclusion

* Extensive intraductal component by the Harvard definition (i.e., more than 25% of the invasive tumor is DCIS and DCIS present in adjacent breast tissue)
* Palpable or radiographically suspicious contralateral axillary, ipsilateral or contralateral supraclavicular, infraclavicular, or internal mammary lymph nodes unless these are histologically confirmed negative
* Patients receiving neoadjuvant chemotherapy
* Patients with distant metastatic disease detected by radiographic imaging; specific studies for systemic imaging should be obtained as directed by localized symptoms or per available NCCN guidelines
* Patients with known BRCA 1/BRCA 2 mutations or those with predicted risk of carrying the mutation by BRCAPRO (44) risk assessment >= 50%
* Diffuse calcifications throughout the breast
* Patients with skin involvement or inflammatory breast cancer
* Patients with Paget's disease of the nipple
* Patients nonepithelial breast malignancies such as lymphoma or sarcoma
* Patients with collagen vascular disorders, specifically systemic lupus erythematosis, scleroderma, or dermatomyositis
* Patients with psychiatric, neurologic, or addictive disorders that would preclude obtaining informed consent
* Other malignancy, except non-melanomatous skin cancer, < 5 years prior to participation in this study
* Patients who are pregnant or lactating, due to potential fetal exposure to radiation and unknown effects of radiation on lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Ipsilateral breast tumor recurrence rates | 5 years after completion of radiation
  Ipsilateral breast 6 months after diagnosis, bilateral annually for 5 years
To determine the cosmetic outcome resulting from breast conserving surgery and breast radiation | at 1 year after radiation

SECONDARY OUTCOMES:
To determine if there are patient factors which limit a patient's suitability to receive breast conserving therapy | 5 years after completion of radiation treatment
Patient satisfaction with the procedure as determined by a questionnaire | at 1 year after radiation
To evaluate wound healing and overall complication rate after radiation | at one year after radiation

CONTACTS AND LOCATIONS:
Overall Officials: William Chen, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - UH-Chagrin Highlands, Orange, Ohio
  - UH-Westlake, Westlake, Ohio

REFERENCES:
- See also: Related Info — http://clinicaltrials.gov/ct2/show/NCT01100489?term=NCT01100489&rank=1